CLINICAL TRIAL: NCT01247363
Title: Safety and Tolerability of Multiple Ascending Doses of LY2608204 in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of LY2608204 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14130; I3P-FW-GKBE (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-11-22; First posted 2010-11-24 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes glucokinase safety
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — globalagliatin; glucokinase activator compound 50

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2608204 (Experimental): Oral capsules of LY2608204 given once daily at a starting dose of 160 milligram (mg), which may be titrated in 3 dose escalations to 240 mg, 320 mg and 400 mg, with a 7-day treatment duration at each dose level for up to 28 days total treatment.
  Interventions: Drug: LY2608204

INTERVENTIONS:
Drug: LY2608204 — Administered orally.
  Other Names: Glucokinase Activator

SUMMARY:
Safety study with multiple oral doses of LY2608204 given to patients with type 2 diabetes. Study subjects will receive once daily doses of LY2608204 for a total treatment duration of up to 28 days. In this study, each patient will receive increasing doses of LY2608204 until reaching the highest dose that they can tolerate.

Continuous glucose monitoring devices will be employed for each patient to monitor for hypoglycemia during study treatment. Dose titration and dose reduction is determined for each individual patient based on their safety and glycemic data.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Type 2 diabetes mellitus (T2DM) who are currently treated with diet/lifestyle measures alone or in combination with anti-diabetic agents, including insulins
* Have fasting blood glucose (FBG) greater than or equal to 160 milligram/deciliter (mg/dL), with a subset of patients with FBG greater than or equal to 190 mg/dL in at least 2 measurements on separate days
* Have a glycated haemoglobin (HbA1c) level of greater than or equal to 8% and less than or equal to 11% at screening
* If female, are not of child-bearing potential due to surgical sterilisation (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause
* Are males or females who are at least 18 years old (for sites outside of Singapore) or at least 21 years old (for sites within Singapore) but no more than 70 years old (for all sites)
* Body mass index (BMI) greater than 18.5 kilogram/square meter (kg/m²) and less than 40.0 kg/m²
* Have clinical laboratory test results within the normal range for the population or investigator site, or with abnormalities deemed clinically insignificant by the investigator
* Have supine systolic blood pressure (SBP) greater than 160 millimeters of mercury (mmHg) and supine diastolic blood pressure (DBP) less than 100 mmHg
* Have venous access sufficient to allow blood sampling as per the protocol
* Are willing and able to comply with requirements for continuous glucose monitoring (CGM)
* Are reliable and willing to make themselves available for the duration of the study and who will abide by the Clinical Research Unit (CRU) policy and procedure and study restrictions. This includes staying in-patient at the CRU for a total duration of up to 31 days
* Have given written informed consent approved by Lilly and the ethical review board governing the site

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device or use of a drug or device other than the study drug used in this study, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have significant history of past or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine (other than diabetes), hematological, or neurological disorders capable of significantly altering the absorption, metabolism or elimination of drugs or of constituting a risk when taking the study drug formulations or interfering with the interpretation of data
* Have a history of a seizure disorder
* A corrected QT interval greater than 450 milliseconds (msec) at screening or any personal history of ventricular tachycardia or unexplained syncope, or other abnormality in the 12-lead Electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have family history of long QT syndrome or family history of sudden unexplained death
* Use medications known to prolong the QT interval.
* Have type 1 diabetes mellitus or a history of ketoacidosis or any other type of diabetes mellitus other than type 2
* Use of any known inducers or inhibitors of CYP3A within 14 days prior to the first dosing with study drug or intended use during the study
* History of a hypoglycemic event with acute mental status alteration that was not preceded by prodromal symptoms recognizable to the patient
* Fasting serum triglycerides greater than 500mg/dl
* Serum creatinine greater than 1.3 mg/dL in women, greater than 1.5 mg/dL in men
* Clinical evidence of active diabetic proliferative retinopathy
* Known clinically significant autonomic neuropathy as evidenced by urinary retention, orthostatic hypotension, diabetic diarrhea or gastroparesis
* Clinically significant coronary events or symptoms within 6 months prior to study entry
* Clinically significant peripheral vascular disease
* Have known allergies to LY2608204 or related compounds
* Evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies/antigen
* Evidence of hepatitis B and/or positive hepatitis B surface antigen (HBsAg)
* Donation or loss of blood equal to or exceeding 450 milliliter (mL) during the 3 months before the first administration of study drug
* Patients who have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females) (1 unit equal to 12 oz or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits) or patients unwilling to stop alcohol consumption 24 hours prior to admission until the completion of each in-patient study period
* Patients who smoke more than 10 cigarettes or other tobacco products per day before study entry. Patients will not be allowed to smoke while in the study Unit
* Have a history of drug or alcohol abuse
* Intended use of over-the counter or prescription medications 7 and 14 days, respectively, prior to dosing. If this situation arises, inclusion of an otherwise suitable volunteer may be at the discretion of the investigator. Use of anti-diabetic medication [metformin, sulphonylureas, glinides, thiazolidinediones, acarbose, DPPIV inhibitors, Byetta (but not liraglutide)] by patients with type 2 diabetes mellitus is acceptable for this study
* Have repeated alanine transaminase levels greater than 2.5 times the upper limit of the reference range at screening, as determined by the central laboratory
* Have previously been enrolled in this clinical study or any other study of LY2608204.

Exclusion Criteria for EU/UK/US Site(s) only --

* Evidence of hepatitis C and/or positive hepatitis C antibodies, at screening
* Use of known drugs of abuse and/or positive findings on urinary drug screening, other than findings consistent with medication prescribed by the patient's physician or over-the-counter medications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miramar, Florida, United States
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2608204: Oral capsules of LY2608204 given once daily at a starting dose of 160 mg, which was titrated in 3 dose escalations to 240 mg, 320 mg and 400 mg, with a 7-day treatment duration at each dose level for up to 28 days total treatment.
Period: Overall Study
Arm/Group | LY2608204
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LY2608204
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2
  White | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Fasting Blood Glucose (FBG) [Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)] | 233.5 (38.61)
Glycated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] — HbA1c is a form of hemoglobin which is measured primarily to identify the average plasma glucose concentration over prolonged periods of time.
  percentage of glycated hemoglobin | 10.48 (0.89)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Adverse Effects
Description: Clinically significant adverse effects refer to any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the investigational product, whether or not related to the medicinal investigational product.
Time Frame: Day 1 through Day 49
Population: Participants who were administered study drug.
Measure: Count of Participants; unit: Participants
Groups:
- 160 mg LY2608204: Oral capsules of LY2608204 given once daily at dose of 160 milligram (mg)
- 240 mg LY2608204: Oral capsules of LY2608204 given once daily at dose of 240 mg
- 320 mg LY2608204: Oral capsules of LY2608204 given once daily at dose of 320 mg
- 400 mg LY2608204: Oral capsules of LY2608204 given once daily at dose of 400 mg
Arm/Group | 160 mg LY2608204 | 240 mg LY2608204 | 320 mg LY2608204 | 400 mg LY2608204
Number analyzed (Participants) | 20 | 20 | 19 | 17
Participants | 9 | 8 | 9 | 8

2. Secondary Outcome: Area Under the Concentration Time Curve (AUC)
Description: AUC for Day 1 is AUC from 0 to 24 hours. AUC for all other days is AUC at a dosing interval.
Time Frame: Predose, 1, 2, 4, 6, 7, 10, 12 and 24 hours Postdose
Population: Participants who were administered study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram.hour/milliliter (ng.hr/mL)
Groups:
- 160 mg LY2608204 Day 1: Oral capsules of LY2608204 given once at dose of 160 milligram (mg)
- 160 mg LY2608204 Day 7: Oral capsules of LY2608204 given once daily at dose of 160 mg
- 240 mg LY2608204 Day 14: Oral capsules of LY2608204 given once daily at dose of 240 mg
- 320 mg LY2608204 Day 21: Oral capsules of LY2608204 given once daily at dose of 320 mg
- 400 mg LY2608204 Day 28: Oral capsules of LY2608204 given once daily at dose of 400 mg
Arm/Group | 160 mg LY2608204 Day 1 | 160 mg LY2608204 Day 7 | 240 mg LY2608204 Day 14 | 320 mg LY2608204 Day 21 | 400 mg LY2608204 Day 28
Number analyzed (Participants) | 20 | 20 | 20 | 19 | 17
nanogram.hour/milliliter (ng.hr/mL) | 1090 (30) | 2780 (30) | 5450 (30) | 8650 (28) | 12100 (35)

3. Secondary Outcome: Maximum Drug Concentration (Cmax)
Time Frame: Predose, 1, 2, 4, 6, 7, 10, 12, 24, 48, 120 and 168 hours Postdose
Population: Participants who were administered study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | 160 mg LY2608204 Day 1 | 160 mg LY2608204 Day 7 | 240 mg LY2608204 Day 14 | 320 mg LY2608204 Day 21 | 400 mg LY2608204 Day 28
Number analyzed (Participants) | 20 | 20 | 20 | 19 | 17
nanogram/milliliter (ng/mL) | 78.7 (33) | 175 (31) | 336 (32) | 515 (30) | 690 (36)

4. Secondary Outcome: Time to Maximum Drug Concentration (Tmax)
Time Frame: Predose, 1, 2, 4, 6, 7, 10, 12, 24, 48, 120 and 168 hours Postdose
Population: Participants who were administered study drug.
Measure: Median (Full Range); unit: hour
Arm/Group | 160 mg LY2608204 Day 1 | 160 mg LY2608204 Day 7 | 240 mg LY2608204 Day 14 | 320 mg LY2608204 Day 21 | 400 mg LY2608204 Day 28
Number analyzed (Participants) | 20 | 20 | 20 | 19 | 17
hour | 6.50 [4.00 to 12.00] | 6.50 [2.00 to 12.00] | 6.00 [4.00 to 10.05] | 6.00 [2.00 to 12.00] | 6.00 [2.00 to 12.00]

5. Secondary Outcome: Number of Hypoglycemic Events
Description: Number of hypoglycemia events with blood glucose concentration <70 milligram/deciliter (mg/dL).
Time Frame: Day 1 through Day 29
Population: Participants who were administered study drug.
Measure: Number; unit: events
Arm/Group | 160 mg LY2608204 | 240 mg LY2608204 | 320 mg LY2608204 | 400 mg LY2608204
Number analyzed (Participants) | 20 | 20 | 19 | 17
events | 0 | 7 | 4 | 0

ADVERSE EVENTS:
Arm/Group | 160 mg LY2608204 | 240 mg LY2608204 | 320 mg LY2608204 | 400 mg LY2608204
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/19 | 0/17
Other Adverse Events (participants affected / at risk) | 9/20 | 8/20 | 9/19 | 8/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 160 mg LY2608204 (N=20) | 240 mg LY2608204 (N=20) | 320 mg LY2608204 (N=19) | 400 mg LY2608204 (N=17)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (3) | 4 (4) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural site reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 1 (1) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (7) | 2 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (10) | 4 (5) | 2 (3) | 2 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days